CLINICAL TRIAL: NCT00592917
Title: OSTPRE-FPS Prevention of Fractures and Falls in Postmenopausal Women With Calcium and Vitamin-D Supplementation - a Randomised Study
Brief Title: OSTPRE-Fracture Prevention Study
Acronym: OSTPRE-FPS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kuopio University Hospital (Other)
Collaborators: University of Eastern Finland (Other); Academy of Finland (Other); Leiras-Nycomed (Unknown)
Responsible Party: Professor Heikki Kroger, Kuopio University Hospital, Dept of Orthopedics, Traumatology and Handsurgery
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KUH5204512; 119/2001
Record Dates: First submitted 2008-01-02; First posted 2008-01-14 (Estimated); Last update posted 2008-01-14 (Estimated); Status verified 2008-01

CONDITIONS: Fractures; Osteoporosis
Keywords: osteoporosis; fractures; risk of fracture; vitamin-D; calcium; falls; bone mineral density; bone metabolism
MeSH Terms: conditions — Fractures, Bone; Osteoporosis | interventions — Calcium Carbonate; Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Ia (Active Comparator): 1718 subjects randomised for active calcium and vitamin-D -intervention, data collection with questionnaires at baseline and end of the study, data of falls and fractures in telephone-interviews annually except Ib (every four months)
  Interventions: Dietary Supplement: calcium carbonate and cholecalciferol
- Ib (Active Comparator): random sample of 292 of 1718 (Ia), data collection by questionnaires mentioned in Ia, data of falls an fractures by telephone interviews every four months, bone density measurements, clinical tests, laboratory sample collections at baseline and end of follow-up as described in study design
  Interventions: Dietary Supplement: calcium carbonate and cholecalciferol
- IIa (No Intervention): 1714 subjects randomised to no intervention group, data collection with questionnaires at baseline and end of the study, data of falls and fractures in telephone-interviews annually except IIb (every four months)
- IIb (No Intervention): random sample of 314 of 1714 (IIa), data collection by questionnaires mentioned in IIa, data of falls an fractures by telephone interviews every four months, bone density measurements, clinical tests, laboratory sample collections at baseline and end of follow-up as described in study design

INTERVENTIONS:
Dietary Supplement: calcium carbonate and cholecalciferol — one tablet (calcium carbonate resembling 500 mg of calcium and 400 IU or 5 micrograms of vitamin-D3, cholecalciferol) twice daily for the whole duration of the study
  Other Names: Calcichew D3 forte (Leiras-Nycomed), ATC-code: A12AX
  Arms: Ia; Ib

SUMMARY:
The purpose of this study is to determine the effect of calcium 1000 mg/d and vitamin-D3 800 IU/d divided in two daily doses on the incidence of falls and fractures, bone mineral density and bone metabolism in postmenopausal women 65-71 years of age.

DETAILED DESCRIPTION:
In aging population osteoporotic fractures in postmenopausal women are a growing problem and a cause of remarkable morbidity, individual suffering and costs. The effect of calcium and vitamin-D in fracture prevention have been tested in elderly patients mostly over 70-75 years of age and results with low dose intervention have been controversial. The aim of this study is to determine the effects of calcium (1000 mg/d) and vitamin-D (800 IU/d) in 65-71 year-old postmenopausal women in a clinical trial on two levels: a) a randomized postal interview trial (n=3432) and b) a randomized clinical trial (n=606). 5407 women of the OSTPRE-cohort received a postal enquiry with questions of health related issues and willingness to participate a calcium and vitamin-D survey. 4706 enquiries were returned. 3432 eligible women were randomised to the active treatment group (n=1718) to receive the intervention and control group (n=1714), that did not receive placebo, they were told to go on as before in terms of calcium or vitamin-D substitution. On the level of the interview trial end point variables, falls and fractures, are collected by telephone interviews annually and on the level of the clinical trial every four months. In clinically examined subset of 606 subjects axial and heel bone mineral density (BMD), heel quantitative ultrasound (QUS) measurement, anthropometric measurements, a comprehensive set of clinical (muscle strength, balance, functional capacity) and laboratory tests (serum calcium, phosphate, AFOS, creatinine, cholesterol, triglycerides, complete blood count, 25-OH-D-vitamin, PTH, osteocalcin and Trap5B and reserve, serum and urine samples) will be performed and food diary will be obtained at baseline and after 3 years follow-up and baseline blood samples will be taken for DNA-analyses.

ELIGIBILITY:
Inclusion Criteria:

* Alive member of the original population based sample (n=14220) of Kuopio Osteoporosis Risk factor and Prevention Study
* Age 65 years or older on 30.11.2002
* Not participating any previous BMD-measurement in OSTPRE
* Living in the province of Kuopio
* Adequately filled baseline enquiry
* Willing to participate calcium and vitamin-D -survey

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 3432 (Actual)
Dates: Start 2002-08; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
fractures | 3 year follow-up

SECONDARY OUTCOMES:
falls | 3 year follow-up
bone mineral density measured by axial DXA, heel pDXA, heel QUS and distal forearm pQCT | 3 year follow-up
markers of bone metabolism | 3 year follow-up
serum vitamin-D levels | 3 year follow-up
serum calcium levels | 3 year follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Heikki P Kroger, Professor, Study Chair — Department of Orthopedics, Traumatology and Hand Surgery, University Hospital of Kuopio; Heikki P Kroger, Professor, Study Director — Department of Orthopedics, Traumatology and Hand Surgery, University Hospital of Kuopio; Marjo Tuppurainen, Professor, Principal Investigator — Department of Gynecology and Obstetrics, University Hospital of Kuopio
Locations (1):
- Bone and Cartilage Research Unit, Clinical Research Centre, University of Kuopio, Kuopio, Finland

REFERENCES:
- [Derived] Karkkainen M, Tuppurainen M, Salovaara K, Sandini L, Rikkonen T, Sirola J, Honkanen R, Jurvelin J, Alhava E, Kroger H. Effect of calcium and vitamin D supplementation on bone mineral density in women aged 65-71 years: a 3-year randomized population-based trial (OSTPRE-FPS). Osteoporos Int. 2010 Dec;21(12):2047-55. doi: 10.1007/s00198-009-1167-8. Epub 2010 Mar 4. PMID 20204604
- [Derived] Salovaara K, Tuppurainen M, Karkkainen M, Rikkonen T, Sandini L, Sirola J, Honkanen R, Alhava E, Kroger H. Effect of vitamin D(3) and calcium on fracture risk in 65- to 71-year-old women: a population-based 3-year randomized, controlled trial--the OSTPRE-FPS. J Bone Miner Res. 2010 Jul;25(7):1487-95. doi: 10.1002/jbmr.48. PMID 20200964